CLINICAL TRIAL: NCT00662922
Title: Does Hypoglycemia Under Intensive Insulin Therapy During Critical Illness Lead to Neurocognitive Dysfunction
Brief Title: Consequences of Hypoglycemia on Intensive Care Unit (ICU) Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principle investigator, Dr. Björn Ellger, Department of Anesthesiology and Intensive Care Medicine
Other Study IDs: 05-AnIt-07
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Critical Illness
Keywords: critical illness; hypoglycemia; neurocognitive dysfunction; intensive insulin therapy
MeSH Terms: conditions — Critical Illness; Hypoglycemia; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with hypoglycemia during intensive care
- 2: patients without hypoglycemia during intensive care

SUMMARY:
Hypoglycemia occurs frequently during intensive blood glucose control in critically ill patients. The incidence of hypoglycaemia is associated with impaired outcome. However, it is hitherto unknown if hypoglycaemia itself predisposes patients to neurological impairment, e.g. cognitive dysfunction, or if it is the underlying medical condition that makes the patient prone to a high risk of hypoglycaemia and, concomitantly, neurocognitive impairment. Therefore we investigate neurocognitive function in patients who had hypoglycemias during their intensive care stay and compare the results to patients without hypoglycaemia whose medical conditions are matched to the hypoglycaemia patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* clinical diagnosis of diabetes mellitus
* brain injury of any kind prior to or upon ICU-admission
* pre-existing mental or psychiatric disorder
* terminal kidney or liver failure prior admission
* drug abuse,
* CPR > 5 min
* HIV
* Lues

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were admitted to the hospital ICU after 2003 are screened for hypoglycemia
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
neurocognitive function | 1 year after ICU discharge

SECONDARY OUTCOMES:
neurocognitive function | 2,3, and 4 years after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Björn Ellger, MD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, University Hospital Muenster
Locations (1):
- Department of Anesthesiology and Intensive Care, University Hospital Münster, Münster, Germany

REFERENCES:
- [Result] Duning T, van den Heuvel I, Dickmann A, Volkert T, Wempe C, Reinholz J, Lohmann H, Freise H, Ellger B. Hypoglycemia aggravates critical illness-induced neurocognitive dysfunction. Diabetes Care. 2010 Mar;33(3):639-44. doi: 10.2337/dc09-1740. Epub 2009 Dec 23. PMID 20032274